CLINICAL TRIAL: NCT02644005
Title: Automated Control of Mechanical Ventilation During General Anaesthesia - A Bicentric Prospective Observational Trial
Brief Title: Automated Control of Mechanical Ventilation During General Anaesthesia
Acronym: AVAS
Status: Completed | Type: Observational
Sponsor: University Hospital Schleswig-Holstein (Other)
Collaborators: Drägerwerk AG & Co. KGaA (Industry)
Responsible Party: Principal Investigator, Norbert Weiler, Prof. Dr. Norbert Weiler, University Hospital Schleswig-Holstein
Other Study IDs: AVAS
Record Dates: First submitted 2015-12-11; First posted 2015-12-31 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Smart Vent Control — Smart Vent Control (SVC) was designed to automatically control the following ventilator settings: mechanical breathing frequency, inspiratory pressure, pressure support, inspiratory time, trigger sensitivity. SVC adjusts the ventilator settings with the aim to keep a patient stable in a target zone (TZ). Numerous predefined TZs exist that can be set according to the current therapeutic situation. All TZs are adoptable by the user for each individual patient and consist of upper and lower limits for tidal volume and for the partial pressure of end-tidal carbon dioxide (PetCO2). Based on these limits, the system classifies the current quality of ventilation, called Classification of Ventilation, and derives new ventilator settings accordingly. SVC is available as a software option on Zeus Infinity Empowered anesthesia machines (Drägerwerk AG & Co. KGAa, Lübeck, Germany) and is approved as a medical product according to 93/42/European Economic Community.

SUMMARY:
Prospective, bicentric observational study to assess a novel system for automated control of mechanical ventilation (Smart Vent Control, SVC) during general anesthesia.

DETAILED DESCRIPTION:
The "Automated control of mechanical ventilation during general anesthesia study (AVAS study) is an international investigator-initiated bicentric observational study investigating the application of Smart Vent Control (SVC) during general anesthesia. The main objective of this study is to describe the application of SVC and to assess its safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Planned elective surgery of the upper limb, lower limb or peripheral vascular surgery in general anesthesia
* Patient is classified as American Society of Anesthesiologists physical status (ASA) I, II or III
* Age ≥ 18 years
* Written consent of the patient for study participation

Exclusion Criteria:

* Mild, moderate or severe acute respiratory distress syndrome (ARDS)[10]
* Known chronic obstructive pulmonary disease Gold stage III or higher
* Two or more of the following organ failures

  * Mild, moderate or severe ARDS
  * Hemodynamic instability: systolic blood pressure < 90 mm Hg, mean arterial pressure < 70 mm Hg or administration of any vasoactive drugs.
  * Acute renal failure: oliguria (urine output < 0.5 ml/kg/h for at least 2 hours despite of adequate management or creatinine increase > 0.5 mg/dl
  * Cerebral failure: loose of consciousness or encephalopathy
* Patient is pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients scheduled for elective surgery in general anesthesia.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-07-07 (Actual); Primary Completion 2019-03-07 (Actual); Study Completion 2019-03-07 (Actual)

PRIMARY OUTCOMES:
Frequency of adverse events. | During artificial ventilation with SVC (up to 8 hours).
  * Severe hypoventilation defined as minute volume lower than 40 ml/kg predicted body weight for longer than 5 minutes
  * Apnea for longer than 90 seconds
  * Hyperventilation defined as PetCO2 lower than 5 mm Hg of the lower target setting for SVC for longer than 5 minutes
  * Hypoventilation defined as PetCO2 higher than 5 mm Hg of the upper target setting for the SVC for longer than 5 minutes
  * Respiratory rate > 35 breaths per minute for longer than 5 minutes
  * Any override or stop of the automated controlled ventilation settings by the anesthesiologist in charge if the settings are clinically not acceptable. Reasons for overriding or stopping the system will be noted.

SECONDARY OUTCOMES:
Frequency of normoventilated, hypoventilated and hyperventilated patients. | During artificial ventilation with SVC (up to 8 hours).
  The responsible anesthesiologist defines a target range for the arterial partial pressure of carbon dioxide (PaCO2_target) before the induction of the general anesthesia and sets up the corresponding endtidal CO2-range in the automated ventilation system. 15 minutes after the begin of the surgical procedure an arterial blood gas analysis will be performed and the PaCO2 will be measured. Then patients will be classified as follows:
  * hypoventilated patient: PaCO2 > (PaCO2_target+5)
  * hyperventilated patient: PaCO2 < (PaCO2_target-5)
  * normoventilated patient: (PaCO2_target-5) ≤ PaCO2 ≤ PaCO2_target+5
Time period between switch from controlled ventilation to augmented ventilation and achievement of stable assisted ventilation of the patient. | During artificial ventilation with SVC (up to 8 hours).
Proportion of time within the target zones for tidal volume and PetCO2 as individually set up for each patient by the user. | During artificial ventilation with SVC (up to 8 hours).
Frequency of alarms. | During artificial ventilation with SVC (up to 8 hours).
Frequency distribution of tidal volume (ml/kg predicted body weight). | During artificial ventilation with SVC (up to 8 hours).
Frequency distribution of inspiratory pressure (mbar). | During artificial ventilation with SVC (up to 8 hours).
Frequency distribution of inspiration time (s). | During artificial ventilation with SVC (up to 8 hours).
Frequency distribution of expiration time (s). | During artificial ventilation with SVC (up to 8 hours).
Frequency distribution of PetCO2 (mmHg). | During artificial ventilation with SVC (up to 8 hours).
Number of re-intubations. | During artificial ventilation with SVC (up to 8 hours).

CONTACTS AND LOCATIONS:
Overall Officials: Norbert Weiler, M.D., Principal Investigator — University Medical Center Schleswig-Holstein, Campus Kiel, Germany, Department of Anesthesiology and Intensive Care Medicine; Christoph Hörmann, M.D., Principal Investigator — University Hospital St. Pölten, Austria, Department of Anesthesiology and Intensive Care Medicine
Locations (2):
- University Hospital St. Pölten, Department of Anesthesiology and Intensive Care Medicine, Sankt Pölten, Austria
- University Medical Center Schleswig-Holstein, Campus Kiel, Department of Anesthesiology and Intensive Care Medicine, Kiel, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schadler D, Miestinger G, Becher T, Frerichs I, Weiler N, Hormann C. Automated control of mechanical ventilation during general anaesthesia: study protocol of a bicentric observational study (AVAS). BMJ Open. 2017 May 10;7(5):e014742. doi: 10.1136/bmjopen-2016-014742. PMID 28495814